CLINICAL TRIAL: NCT03695094
Title: A Multicenter, Open-label, Parallel-group Study in Study Participants With Epilepsy, to Evaluate the Effect of Oxcarbazepine on the Pharmacokinetics, Safety, and Tolerability of Padsevonil
Brief Title: A Study in Participants With Epilepsy, to Evaluate the Pharmacokinetics, Safety and Tolerability of Oxcarbazepine on Padsevonil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP0070; 2018-001941-16 (EudraCT Number)
Record Dates: First submitted 2018-09-14; First posted 2018-10-03 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Phase 1; padsevonil
MeSH Terms: conditions — Epilepsy | interventions — padsevonil; Oxcarbazepine; Levetiracetam; Lamotrigine; brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 (Inducers): Study participants on stable therapy with oxcarbazepine (OXC) either as monotherapy or adjunctive to levetiracetam (LEV), lamotrigine (LTG), or brivaracetam (BRV). OXC may be used as monotherapy or in combination with 1 or more of LEV, LTG, or BRV. Padsevonil (PSL) will be dosed to steady state and the effect of background therapy on PSL pharmacokinetics will be assessed at steady state.
  Interventions: Drug: Padsevonil; Drug: Oxcarbazepine; Drug: Levetiracetam; Drug: Lamotrigine; Drug: Brivaracetam
- Cohort 2 (Experimental): Cohort 2 (Neutral): Study participants on stable therapy with lamotrigine (LTG), levetiracetam (LEV), or brivaracetam (BRV). LTG or LEV may be used as monotherapy or in combination with each other. BRV may only be used in combination with LTG. LTG or LEV may be used as monotherapy or in combination with each other. BRV may only be used in combination with LTG. Padsevonil (PSL) will be dosed to steady state (4.5 days) and the effect of background therapy on PSL pharmacokinetics will be assessed at steady state.
  Interventions: Drug: Padsevonil; Drug: Levetiracetam; Drug: Lamotrigine; Drug: Brivaracetam

INTERVENTIONS:
Drug: Padsevonil — Padsevonil (PSL) will be dosed to steady state and the effect of background therapies on pharmacokinetics will be assessed
  Other Names: PSL; UCB0942
Drug: Oxcarbazepine — Concomitant administration of oxcarbazepine (OXC) at therapeutic dosage
  Other Names: OXC
  Arms: Cohort 1
Drug: Levetiracetam — Concomitant administration of levetiracetam (LEV) at therapeutic dosage
  Other Names: LEV
Drug: Lamotrigine — Concomitant administration of lamotrigine (LTG) at therapeutic dosage
  Other Names: LTG
Drug: Brivaracetam — Concomitant administration of brivaracetam (BRV) at therapeutic dosage
  Other Names: BRV

SUMMARY:
The purpose of the study is to evaluate the effect of stable coadministered oxcarbazepine (OXC), on the pharmacokinetics (PK), safety, tolerability of padsevonil (PSL) and the plasma PK of PSL metabolites, UCB1431322-000 and UCB1447499-000, in study participants with epilepsy compared with study participants co-medicated with stable doses of levetiracetam (LEV), lamotrigine (LTG) or brivaracetam (BRV) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Study participant is male or female between 18 to 64 years of age, inclusive, with a diagnosis of epilepsy according to the International League Against Epilepsy (ILAE) classification
* Study participant is currently treated for epilepsy with stable doses of the following for at least 3 months:

  1. Inducers Group: Oxcarbazepine (OXC) (at least 1200 mg/day as monotherapy or in combination with brivaracetam (BRV) [up to 200 mg/day], levetiracetam (LEV) [at least 1 g/day] or lamotrigine (LTG) [at least 150 mg/day]); or
  2. Neutral (control) Group: LTG (at least 150 mg/day monotherapy or adjunctive to LEV or BRV), LEV (at least 1 g/day monotherapy or adjunctive to LTG), or BRV (up to 200 mg/day adjunctive to LTG)
* Study participant in the Inducers Group is taking OXC and has a trough OXC metabolite Mono Hydroxy Derivate (MHD) plasma level in the target range (≥12.0 to ≤35.0 mcg/mL)
* Study participant has clinical laboratory test results within the local reference ranges or values are considered as not clinically relevant by the Investigator and approved by the UCB Study Physician
* Study participant has a body mass index (BMI) of 18 to 35 kg/m², inclusive, with a body weight of at least 50 kg (male) or 45 kg (female)
* Female study participant has a negative serum pregnancy test at the Screening Visit and agrees to use an efficient form of contraception for the duration of the study (unless menopausal [defined as no menses for 12 months without an alternative medical cause]; a high follicle-stimulating hormone level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy). -Male study participant agrees that, during the study period, when having sexual intercourse with a woman of childbearing potential, he will use an efficient barrier contraceptive (condom plus spermicide) AND that the respective partner will use an additional efficient contraceptive method (eg, oral pills, intrauterine device, intrauterine hormone-releasing systems, or diaphragm, and spermicide)

Exclusion Criteria:

* Study participant has participated in another study of an investigational medication (or a medical device) within the last 3 months before screening (or 5 half-lives, whichever is longer) or is currently participating in another study of an investigational medication (or a medical device)
* Study participant has a known hypersensitivity to any components of the IMP as stated in this protocol
* Study participant has any medical condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Study participant has a history of status epilepticus during the last year
* Study participant has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline
* Study participant has received any prescription or nonprescription medicines, including enzyme inhibitors or inducers, over the counter (OTC) remedies, herbal and dietary supplements (including St. John's Wort), or vitamins up to 2 weeks or 5 half-lives of the respective drug (whichever is longer) before the first administration of IMP and during the clinical part of the study, unless required to treat an Adverse event (AE). This does not include allowed antiepileptic drugs (AEDs) per the protocol, oral contraceptives not exceeding 30 μg ethinyl estradiol or postmenopausal hormone replacement therapy or implants, patches, or IUDs/IUSs delivering progesterone (for female study participants)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (2):
- Up0070 101, Sofia, Bulgaria
- Up0070 401, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chanteux H, MacPherson M, Kramer H, Otoul C, Okagaki T, Rospo C, De Bruyn S, Watling M, Bani M, Sciberras D. Overview of preclinical and clinical studies investigating pharmacokinetics and drug-drug interactions of padsevonil. Expert Opin Drug Metab Toxicol. 2024 Aug;20(8):841-855. doi: 10.1080/17425255.2024.2373108. Epub 2024 Jul 9. PMID 38932723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in September 2018 and concluded in May 2019.
Pre-assignment Details: The study included a Screening Period (Day -28 to Day -2), a Baseline Visit (Day -1), a Treatment Period (Day 1 to Day 12) and a Safety Follow-Up Period Day (13 to Day 20±1).
  Participant Flow refers to the Full Analysis Set.
Groups:
- Group 1 (Inducers): Participants were on stable therapy with oxcarbazepine (OXC), at least 1200 milligrams per day (mg/day), which could be used as monotherapy or adjunctive to 1 or more of levetiracetam (LEV), lamotrigine (LTG), or brivaracetam (BRV). Padsevonil (PSL) was dosed to steady state (4.5 days) and the effect of background therapy on PSL pharmacokinetics (PK) was assessed at steady state.
- Group 2 (Neutral [Control]): Participants were on stable therapy with LTG (at least 150 mg/day monotherapy or adjunctive to LEV or BRV), LEV (at least 1 g/day monotherapy or adjunctive to LTG), or BRV (up to 200 mg/day adjunctive to LTG). Padsevonil (PSL) was dosed to steady state (4.5 days) and the effect of background therapy on PSL pharmacokinetics (PK) was assessed at steady state.
Period: Overall Study
Arm/Group | Group 1 (Inducers) | Group 2 (Neutral [Control])
Started | 16 | 15
Completed | 14 | 14
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Full Analysis Set (FAS) which consisted of all study participants who signed the Informed Consent Form (ICF) and received at least 1 dose of investigational medicinal product (padsevonil).
Arm/Group | Group 1 (Inducers) | Group 2 (Neutral [Control]) | Total Title
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.1) | 33.6 (10.4) | 37.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 14 | 30
  Other or mixed | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Observed Plasma Concentration (Cmax) of Padsevonil (PSL) During the Study
Description: The Cmax for Padsevonil in plasma was expressed in nanograms per milliliter (ng/mL).
Time Frame: Blood samples were taken on Day 1 through Day 12, prior to the morning dose of PSL, at Day 13 prior to unit discharge and at Day 8 at pre-defined time points up to 12 hours post-dose
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) was a subset of the Full Analysis Set (FAS), consisting of study participants who had no important protocol deviations affecting the PK parameters and for whom a sufficient number of samples were available to determine at least 1 PK parameter.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Group 1 (Inducers) (PK-PPS): Participants were on stable therapy OXC, at least 1200 mg/day, which could be used as monotherapy or adjunctive to 1 or more of LEV, LTG, or BRV. Padsevonil (PSL) was dosed to steady state (4.5 days) and the effect of background therapy on PSL pharmacokinetics (PK) was assessed at steady state. Participants formed the Pharmacokinetic Per-Protocol Set (PK-PPS).
- Group 2 (Neutral [Control]) (PK-PPS): Participants were on stable therapy with LTG (at least 150 mg/day monotherapy or adjunctive to LEV or BRV), LEV (at least 1 g/day monotherapy or adjunctive to LTG), or BRV (up to 200 mg/day adjunctive to LTG). Padsevonil (PSL) was dosed to steady state (4.5 days) and the effect of background therapy on PSL pharmacokinetics (PK) was assessed at steady state. Participants formed the PK-PPS.
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
ng/mL | 1210 [1010 to 1450] | 1670 [1390 to 2000]
Statistical Analysis 1: Comparison: Group 1 (Inducers) (PK-PPS) vs Group 2 (Neutral [Control]) (PK-PPS); The analysis of variance model (ANOVA) included the fixed effects of treatment group. The natural logs were taken of the dependent variables and were back-transformed after the analysis. The geometric mean ratio and the respective 90% confidence interval (CI) was derived for the Inducers group vs the Neutral-control group from the ANOVA model using least-squares means difference; Test type: Other; ANOVA; Geometric mean ratio = 0.725, 90% CI 2-sided [0.586 to 0.896]

2. Primary Outcome: The Time to Reach Maximum Concentration (Tmax) for Padsevonil During the Study
Description: The tmax for Padsevonil in plasma was expressed in hours (hr).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
hr | 1.500 [1.00 to 4.00] | 2.000 [0.500 to 4.00]

3. Primary Outcome: The Area Under the Plasma Concentration Time Curve (AUCtau) Over a Dosing Interval for PSL
Description: The AUCtau for Padsevonil in plasma was expressed in hours times nanograms per milliliter (hr*ng/mL).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
hr*ng/mL | 5301 [4350 to 6460] | 8339 [6850 to 10200]
Statistical Analysis 1: Comparison: Group 1 (Inducers) (PK-PPS) vs Group 2 (Neutral [Control]) (PK-PPS); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Geometric mean ratio = 0.636, 90% CI 2-sided [0.504 to 0.801]

4. Primary Outcome: The Apparent Total Plasma Clearance at Steady-state (CL/Fss) for PSL During the Study
Description: The CL/Fss for Padsevonil in plasma was expressed in liters per hour (L/hr). Geometric Means and Coefficients of Variation (CVs) were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
L/hr | 75.44 (34.8) | 47.94 (39.3)

5. Secondary Outcome: Trough Plasma Concentration of Mono Hydroxy Derivate (MHD) in the Inducers Group Before, During and After Dosing to Steady State With PSL
Description: The trough plasma concentration of MHD with PSL was expressed in micrograms per milliliter (µg/mL).
  Geometric Means and Coefficients of Variation (CVs) were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: Trough plasma samples were taken prior to the morning dose of OXC on Day -1, Day 1 through Day 20 (+/-1)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group 1 (Inducers) (PK-PPS)
Number analyzed (Participants) | 14
µg/mL
  Day 1 | 14.9 (14.5)
  Day 2 | 14.0 (21.6)
  Day 3 | 14.9 (17.0)
  Day 4 | 15.5 (16.0)
  Day 5 | 15.2 (17.5)
  Day 6 | 15.4 (18.1)
  Day 7 | 15.4 (17.0)
  Day 8 | 16.3 (16.1)
  Day 9: number analyzed (Participants) | 13
  Day 9 | 15.4 (13.2)
  Day 10 | 15.5 (13.8)
  Day 11 | 15.4 (18.6)
  Day 12 | 13.8 (20.9)
  Day 13: number analyzed (Participants) | 13
  Day 13 | 11.3 (46.4)

6. Secondary Outcome: The Maximum Observed Plasma Concentration (Cmax) for UCB1431322-000 During the Study
Description: The Cmax for UCB1431322-000 in plasma was expressed in nanograms per milliliter (ng/mL).
  Geometric Means and Coefficients of Variation (CVs) were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
ng/mL | 1753 (21.7) | 1700 (29.4)

7. Secondary Outcome: The Time to Reach Maximum Concentration (Tmax) for UCB1431322-000 During the Study
Description: The tmax for UCB1431322-000 in plasma was expressed in hours (hr).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
hr | 3.500 [1.00 to 4.00] | 3.500 [1.00 to 4.00]

8. Secondary Outcome: The Area Under the Curve (AUCtau) Over a Dosing Interval for UCB1431322-000 During the Study
Description: The AUCtau for UCB1431322-000 in plasma in was expressed in hours times nanograms per milliliter (hr*ng/mL).
  Geometric Means and Coefficients of Variation (CVs) were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
hr*ng/mL | 11720 (21.3) | 11200 (30.7)

9. Secondary Outcome: The Ratio of PSL Metabolite UCB1431322-000 to PSL Based on the Area Under the Curve (AUCtau) During the Study
Description: Metabolite-to-Parent Ratios were corrected for differences in molecular weight. Geometric Means and Coefficients of Variation (CVs) were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
ratio | 2.283 (22.4) | 1.386 (48.2)

10. Secondary Outcome: The Maximum Observed Plasma Concentration (Cmax) for UCB1447499-000 During the Study
Description: The Cmax for UCB1447499-000 in plasma was expressed in ng/mL. Geometric Means and Coefficients of Variation (CVs) were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
ng/mL | 380.1 (37.8) | 307.2 (32.6)

11. Secondary Outcome: The Time to Reach Maximum Concentration (Tmax) for UCB1447499-000 During the Study
Description: The tmax for UCB1447499-000 in plasma was expressed in hr.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
hr | 2.000 [1.00 to 4.00] | 2.000 [1.50 to 4.00]

12. Secondary Outcome: The Area Under the Curve (AUCtau) Over a Dosing Interval for UCB1447499-000 During the Study
Description: The AUCtau for UCB1447499-000 in plasma was expressed in hr*ng/mL. Geometric Means and Coefficients of Variation (CVs) were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
hr*ng/mL | 1854 (29.0) | 1678 (28.2)

13. Secondary Outcome: The Ratio of PSL Metabolite UCB1447499-000 to PSL Based on the Area Under the Curve (AUCtau)
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Group 1 (Inducers) (PK-PPS) | Group 2 (Neutral [Control]) (PK-PPS)
Number analyzed (Participants) | 14 | 14
ratio | 0.3492 (32.8) | 0.2011 (45.7)

14. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During the Study
Description: An AE was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From screening (Day -28 to Day -2) up to end of study (EOS) visit day 20 (+/-1)
Population: The Full Analysis Set (FAS) consisted of all study participants who signed the ICF and received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Groups:
- Group 1 (Inducers) (FAS): Participants were on stable therapy with oxcarbazepine (OXC), at least 1200 mg/day, which could be used as monotherapy or adjunctive to 1 or more of levetiracetam (LEV), lamotrigine (LTG), or brivaracetam (BRV). Padsevonil (PSL) was dosed to steady state (4.5 days) and the effect of background therapy on PSL pharmacokinetics (PK) was assessed at steady state. Participants formed the Full Analysis Set (FAS).
- Group 2 (Neutral [Control]) (FAS): Participants were on stable therapy with LTG (at least 150 mg/day monotherapy or adjunctive to LEV or BRV), LEV (at least 1 g/day monotherapy or adjunctive to LTG), or BRV (up to 200 mg/day adjunctive to LTG). Padsevonil (PSL) was dosed to steady state (4.5 days) and the effect of background therapy on PSL pharmacokinetics (PK) was assessed at steady state. Participants formed the FAS.
Arm/Group | Group 1 (Inducers) (FAS) | Group 2 (Neutral [Control]) (FAS)
Number analyzed (Participants) | 16 | 15
percentage of participants | 100 | 100

15. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE) During the Study
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required in patient hospitalization or prolongation of existing hospitalization, was a congenital anomaly or birth defect, was an infection that requires treatment parenteral antibiotics or other important medical events which based on medical or scientific judgement could jeopardize the patients, or could require medical or surgical intervention to prevent any of the above.
Time Frame: From screening (Day -28 to Day -2) up to end of study (EOS) visit day 20 (+/-1)
Population: The Full Analysis Set (FAS) consisted of all study participants who signed the ICF and received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 (Inducers) (FAS) | Group 2 (Neutral [Control]) (FAS)
Number analyzed (Participants) | 16 | 15
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse events (TEAEs) were collected from the Baseline Visit (Day -1) until the Safety Follow-Up Period (Day 20±1).
Description: Only TEAEs occurring above the reporting threshold of 5% of participants in any treatment group are included in this summary.
Arm/Group | Group 1 (Inducers) (FAS) | Group 2 (Neutral [Control]) (FAS)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 16/16 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Inducers) (FAS) (N=16) | Group 2 (Neutral [Control]) (FAS) (N=15)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 1 (3)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (9)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 6 (18)
Feeling drunk (General disorders) | 0 (0) | 3 (4)
Gait disturbance (General disorders) | 1 (1) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Crying (General disorders) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Sluggishness (General disorders) | 0 (0) | 1 (2)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 1 (1)
Blood calcium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 12 (13) | 12 (53)
Dizziness (Nervous system disorders) | 9 (18) | 10 (62)
Headache (Nervous system disorders) | 8 (15) | 9 (23)
Sudden onset of sleep (Nervous system disorders) | 0 (0) | 8 (36)
Amnesia (Nervous system disorders) | 1 (2) | 4 (5)
Disturbance in attention (Nervous system disorders) | 0 (0) | 4 (8)
Focal dyscognitive seizures (Nervous system disorders) | 1 (4) | 3 (3)
Head discomfort (Nervous system disorders) | 0 (0) | 2 (3)
Anterograde amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (2)
Dysgraphia (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Slow response to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Stupor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (8)
Disorientation (Psychiatric disorders) | 2 (2) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 2 (3)
Depressed mood (Psychiatric disorders) | 0 (0) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 1 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03695094/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT03695094/SAP_001.pdf